CLINICAL TRIAL: NCT05078203
Title: Acute Exercise and Cognitive Function: Examining the Role of Weight Status and Exercise-Induced Myokines
Brief Title: Acute Cognition and Exercise
Acronym: ACE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Urbana-Champaign (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: ACE
Record Dates: First submitted 2021-10-01; First posted 2021-10-14 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Obesity
Keywords: Myokine; Cognition; CTSB; BDNF; Exercise
MeSH Terms: conditions — Obesity; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: 18 adults with healthy weight (BMI 18.5-25.0kg/m2) and 18 adults with obesity (BMI 30.0kg/m2) will be asked to complete a counter-balanced crossover trial. After initial baseline testing, participants will be asked to complete either an acute exercise bout or sedentary control session in a counter-balanced order.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise (Experimental): 36 minutes of exercise
  Interventions: Behavioral: Exercise
- Rest (Placebo Comparator): 36 minutes of rest
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — 36 minutes of Exercise

SUMMARY:
The central hypothesis is that, while both groups will benefit from the exercise session, participants with obesity will exhibit greater gains in cognitive control, relative to healthy weight adults. Additionally, it is anticipated that the benefits of a single bout of exercise for cognitive control will be mediated by changes in exercise-induced myokines. These hypotheses will be tested by accomplishing three aims:

Aim 1: Elucidate the changes in cognitive control following an acute bout of exercise, relative to a sedentary condition, in persons with and without obesity.

Aim 2: To examine the effect of a single bout of exercise, relative to a sedentary condition, on myokines known to have neuroprotective effects i.e., BDNF and CTSB in both healthy weight and individuals with obesity.

Aim 3: To link changes in exercise-induced myokines (i.e., BDNF and CTSB) to changes in cognitive function, following a single bout of exercise.

DETAILED DESCRIPTION:
18 adults with healthy weight (BMI 18.5-25.0kg/m2) and 18 adults with obesity (BMI 30.0kg/m2) will be asked to complete a counter-balanced crossover trial. After initial baseline testing, participants will be asked to complete either an acute exercise bout or sedentary control session in a counter-balanced order. A cognitive testing battery accompanied by an electroencephalogram (EEG) will be administered following each session. Blood samples will be collected prior to, during, and following each throughout each testing condition.

ELIGIBILITY:
Inclusion Criteria:

* Between ages 18 and 35
* No prior diagnosis of neurological disorders (e.g., autism spectrum disorder)
* No prior diagnosis of metabolic disease (e.g., diabetes, cardiovascular disease)
* No physical disability that would preclude the participant from completing a VO2max test
* Corrected vision (based on the minimal 20/20 standard needed to complete cognitive tasks)
* Not pregnant
* BMI between 18.5 and 25.0 kg/m2, or BMI greater than 30.0 kg/m2
* Readiness for exercise (determined through PAR-Q)

Exclusion Criteria:

* <18 years and >35 years
* Diagnosis of neurological disorders (e.g., autism spectrum disorder)
* Diagnosis of metabolic disease (e.g., diabetes, cardiovascular disease)
* Physical disability that would preclude the participant from completing a VO2max test
* Lack of corrected vision (based on the minimal 20/20 standard needed to complete cognitive tasks)
* Pregnancy
* BMI less than 18.5 kg/m2 or BMI greater than 25.0 but less than 30.0 kg/m2

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2021-09-02 (Actual); Primary Completion 2022-04-28 (Actual); Study Completion 2022-04-28 (Actual)

PRIMARY OUTCOMES:
Circulating Cathepsin B (CTSB) Myokine | 3 hours
  Changes in peripheral myokine concentration
Attentional Inhibition Accuracy | 3 hours
  Behavioral performance measured as accuracy (%) during Flanker task
Attentional Inhibition Reaction Time | 3 hours
  Behavioral performance measured as response time (ms) during Flanker task
Attentional Resource Allocation | 3 hours
  Changes in P3 event related potential amplitude (microvolts) using a computerized flanker task
Attentional Processing Speed | 3 hours
  Changes in P3 event related potential latency (ms) using a computerized flanker task
Relational Memory | 3 hours
  Accuracy during a spatial reconstruction task

SECONDARY OUTCOMES:
Brain derived neurotrophic factor (BDNF) | 3 hours
  Changes in peripheral BDNF concentration

CONTACTS AND LOCATIONS:
Locations (1):
- University of Illinois at Urbana-Champaign, Urbana, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided